CLINICAL TRIAL: NCT01873469
Title: Observational Study of Impact of [11C]-Methionine PET/MRI as a Tool for Individual Tailoring Postoperative Radiochemotherapy for Patients With Glioblastoma Multiforme
Brief Title: Impact of [11C]-Methionine PET/MRI for Individual Tailoring Postoperative Radiochemotherapy for Glioblastoma Multiforme
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Mechthild Krause, PD Dr. med., Technische Universität Dresden
Other Study IDs: STR-PETra-2013
Record Dates: First submitted 2013-06-04; First posted 2013-06-10 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma multiforme; radiotherapy
MeSH Terms: conditions — Glioblastoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh tumour pieces, blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiochemotherapy: glioblastoma patients with indication to radiochemotherapy
  Interventions: Radiation: Radiochemotherapy

INTERVENTIONS:
Radiation: Radiochemotherapy — postoperative radiochemotherapy 60 Gy/ Temozolomide

SUMMARY:
Local recurrence is a major problem of clinical treatment of glioblastoma multiforme (GBM). Today a very sensitive imaging method to detect glioblastoma is [11C]MET Positron emission tomography (PET), where in some patients also tumour manifestations can be detected that are not visible in MRI investigations.

The aim of the study is to investigate the association of high [11C]MET tracer uptake before postoperative radiochemotherapy and concurrent temozolomide (TMZ) with time to recurrence in patients with glioblastoma multiforme. Also site of recurrence will be correlated with the [11C]MET imaging before and early during radiochemotherapy. All imaging information will be included in treatment planning or treatment decisions.

The study provides a basis for later radiation dose escalation trials on the base of [11C]MET imaging.

DETAILED DESCRIPTION:
The current study aims to investigate the association of high [11C]MET tracer uptake before postoperative radiochemotherapy and concurrent temozolomide (TMZ) with time to recurrence in patients with glioblastoma multiforme (GBM).

[11C]MET-PET is expected to provide diagnostic (quantitative and spatial information) as well as prognostic information, to monitor treatment, to help stratification of patients for radiotherapeutic interventions such as dose-painting in order to optimize clinical applications and potentially improve the treatment outcome.

This study aims to provide the basis (e.g. optimal threshold value, sensitivity, specificity of MET uptake) for later intervention trials for treatment intensification, e.g. proton boost irradiation based on specific biomarkers.

The trial is a one-arm single-center, non-randomized observational (biomarker) study. After resection or biopsy, patients with newly diagnosed glioblastoma multiforme will receive a [11C]MET-PET/MRI scan before start of concurrent radiochemotherapy (~1-4 weeks after surgery). A fusion with the planning CT for irradiation treatment planning will be performed. Postoperative radiotherapy will be applied in daily fractions of 2 Gy given 5 days per week for 6 weeks, for a total dose of 60 Gy (50 Gy and a boost of 10 Gy), with concomitant administration of daily Temozolomide (75 mg/m2 p.o.) from the 1st day to the last day of radiotherapy. Follow up with [11C]MET-PET/MRI will be performed every 3 months until recurrence or until death of the patient.

The uptake of [11C]MET-PET (as standard uptake value - SUV) in tumour and in normal contralateral grey matter before start of concurrent radiochemotherapy will be determined. For each tumour, the ratio between tracer uptake in the tumor and contralateral gray matter will be calculated (lesion-to-gray matter ratio [l/g]).

Primary end point will be time to recurrence (TTR) as function of [11C]MET uptake before chemoradiotherapy. Secondary endpoints will be overall survival; toxicity; C-Index/ROC curve (sensitivity, specificity, optimal threshold for normal/tumour tissue index), necrosis rate; site of recurrence.

The primary analysis will use the Cox proportional hazard model to establish the linear association between [11C]-MET and time-to-recurrence using a one-sided alpha = 0.1.

Parallel translational studies with orthotopic GBM xenografts (generated from the patients material in the trial) in nude mice will be performed in our laboratory to evaluate [11C]MET-PET as a tool for tailoring high precision radiotherapy. Histological, biological and genetic studies are planned to validate the imaging finding and to explore the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed newly diagnosed glioblastoma multiforme
* macroscopic total tumour resection or biopsy
* indication for combined radiochemotherapy with temozolomide
* patients are allowed to take part in other clinical trials at the same time
* beginning of radiochemotherapy no later than 7 weeks after surgery
* Karnofsky Performance Score ≥ 60, ECOG ≤2
* women with childbearing potential, (and men) adequate contraception
* ability of subject to understand character and individual consequences of the clinical trial
* written informed consent

Exclusion Criteria:

* previous radiotherapy of the brain or chemotherapy with TMZ other than during the radiochemotherapy
* time interval of > 7 weeks after surgery and beginning of radiochemotherapy
* patients who are not suitable for radiochemotherapy
* known other malignant disease that impacts prognosis of the patient and/or is likely to require treatment interfering with study therapy
* pregnant or lactating women
* patients with non-MRI compatible metal implants, pacemaker or non-MRI compatible external automatic defibrillators, insulin pumps, neurostimulators, cochlear implants
* Claustrophobic patients
* refusal of the patients to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of glioblastoma multiforme
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-07; Primary Completion 2017-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Time to recurrence as function of [11C]MET uptake before postoperative radiochemotherapy | participants will be followed until tumour recurrence, an expected average of 7 months

SECONDARY OUTCOMES:
overall survival | expected average 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, MD, Study Chair — Dresden University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology; and DKTK partner site Dresden
Locations (1):
- Dresden University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Oncology; and DKTK partner site Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No